CLINICAL TRIAL: NCT03553160
Title: Caloric Titration Method of Weight Loss and Maintenance in the Cornell Community: A Longitudinal Analysis of Psychological Factors
Brief Title: Caloric Titration Method of Weight Loss and Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1007001556
Record Dates: First submitted 2018-05-04; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Frequent Self-Weighing (Other): Study examined the effectiveness of daily self-weighing to prevent age related weight gain.
  Interventions: Other: Frequent Self-Weighing

INTERVENTIONS:
Other: Frequent Self-Weighing — Were given scales to weigh themselves daily. Change in weight was measured at the beginning and end of the two year observation period.
  Other Names: Daily weighing

SUMMARY:
Study examined the effectiveness of daily self-weighing to prevent age related weight gain.

DETAILED DESCRIPTION:
Were given scales to weigh themselves daily. Change in weight was measured at the beginning and end of the two year observation period.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* not pregnant
* not trying to gain or lose weight

Exclusion Criteria:

* diabetes
* history of an eating disorder
* Body Mass Index (BMI) greater than 27.0 kg/m2.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-08-16 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2012-09-01 (Actual)

PRIMARY OUTCOMES:
Prevention of age related weight gain by weighing daily | 2 years
  By weighing oneself daily and seeing a graph of their weight on the scale, the participants will be able to prevent gaining weight over a two year period

CONTACTS AND LOCATIONS:
Locations (1):
- Dorms or student houseing, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: No
We have no plan to share the results, but will gladly do if required.